CLINICAL TRIAL: NCT00988351
Title: Portable Monitoring and APAP Treatment for Diagnosis and Treatment of OSA
Brief Title: Continuous Positive Airway Pressure (PAP) Titration and Treatment Versus Auto-adjusting PAP Treatment for Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Florida Foundation for Research and Education (Other)
Responsible Party: Principal Investigator, Richard Berry, Professor of Medicine University of Florida, North Florida Foundation for Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFIRB#384-09
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; positive airway pressure; portable monitoring; auto positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSG CPAP titration then CPAP treatment (Active Comparator): Patients diagnosed with sleep apnea will have a continuous positive airway pressure (CPAP) titration with polysomnography (PSG) followed by continuous positive airway pressure (CPAP) Treatment
  Interventions: Device: Continuous positive airway pressure
- Auto-Adjusting Positive Airway Pressure (Active Comparator): Following diagnosis of obstructive sleep apnea patients will be have auto-adjusting positive airway pressure treatment without a titration.
  Interventions: Device: Auto-adjusting positive airway pressure treatment

INTERVENTIONS:
Device: Continuous positive airway pressure — continuous positive airway pressure determined by polysomnography titration
  Other Names: CPAP
  Arms: PSG CPAP titration then CPAP treatment
Device: Auto-adjusting positive airway pressure treatment — Pressure range 4-18 centimeters of water (cm H2O)
  Other Names: AutoCPAP; APAP
  Arms: Auto-Adjusting Positive Airway Pressure

SUMMARY:
The purpose of this randomized prospective study is to compare the efficacy of two approaches to initiate Positive Airway Pressure (PAP) treatment in patients diagnosed as having obstructive sleep apnea (OSA) by portable monitoring (PM) (limited sleep study). One pathway involves attended Continuous Positive Airway Pressure (CPAP) titration by PSG (full attended sleep study) followed by CPAP treatment. The other pathway involves treatment with auto-adjusting positive airway pressure (APAP)(without a titration). Study Aims: Compare PAP adherence, improvement in subjective sleepiness (Epworth Sleepiness Scale), reaction time (Psychomotor vigilance test), quality of life by the Functional Outcomes of Sleep Questionnaire (FOSQ), and PAP satisfaction (PAP satisfaction questionnaire) between the two study arms.

DETAILED DESCRIPTION:
RESEARCH PLAN: All patients being evaluated for possible OSA are required to attend a Sleep Education and Evaluation Class before having a sleep study. At this class they receive information on sleep apnea, PAP treatment, and the types of sleep studies. They also complete a sleep questionnaire to identify co-existing sleep disorders and important co-morbid medical conditions. Screening of the sleep questionnaire and the patient's medical record is part of routine care to identify patients needing a diagnostic PSG and/or an attended titration. At the end of the class, participation in the current study will be offered the patients. Those signifying interest in being part of the research study and meeting inclusion and exclusion criteria will be contacted to participate in the study. Once they sign an informed consent they will be randomized to one of the two clinical pathways.

METHODS: Study visits:

Before informed consent (routine clinical care)

1. Sleep Education and Evaluation Class (education about OSA, sleep studies, and OSA treatment). Patients complete screening sleep and medical history questionnaires.
2. Determination of patient interest in participating in the current study and review of inclusion/exclusion criteria

After informed consent

1. PM study
2. Randomization if the Portable monitoring (PM) study is diagnostic of OSA. If not, the patient will be offered a diagnostic PSG. If this is positive, they will have APAP treatment. If both the PM and PSG are negative for OSA the patient exits the study but will be followed in sleep clinic.
3. PSG for CPAP titration (PSG arm only).
4. CPAP/APAP setup - patient fills out Epworth Sleepiness Scale (ESS) and Functional Outcomes of Sleep Questionnaire (FOSQ). The same Research coordinator/Respiratory therapist will setup the units, fit masks, and instruct the patients on the use of their device. Patients being treated with CPAP or APAP will be in separate classes.
5. Telephone contact within 7 days of setup with early intervention for PAP problems if needed.
6. Clinic visit 6 weeks after starting treatment: download objective adherence, ESS, FOSQ, and PAP satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* OSA, Apnea-hypopnea index > 5/hour

Exclusion Criteria:

* Prior CPAP
* Uncontrolled Depression
* Moderate to Severe chronic obstructive pulmonary disease (COPD)
* Hypoventilation
* Average estimated nightly total sleep time < 4 hours
* Shift work
* Unstable depression
* Upper airway surgery
* Uncontrolled Restless legs syndrome (RLS), narcolepsy
* Use of supplemental oxygen
* Severe congestive heart failure
* Use of nightly potent narcotics
* Severe obesity (BMI > 40)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Berry, MD, Principal Investigator — University of Florida/Malcom Randall VAMC
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Started | 78 | 78
CPAP Titration | 78 (8 declined CPAP treatment) | 78 (no titration needed)
PAP Setup | 70 (CPAP treatment started) | 78 (APAP treatment started)
Clinic Visit | 64 (6 lost to follow-up or no show for clinic) | 69 (9 lost to follow-up or no show for clinic)
Using CPAP or APAP | 59 (5 not using CPAP (use < 1/2 hour per night)) | 66 (3 not using APAP (less than 1/2 hour per night))
Completed | 59 | 66
Not Completed | 19 | 12
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Lost to Follow-up | 6 | 9
Not completed — not using CPAP | 5 | 3

BASELINE CHARACTERISTICS:
Population: Apnea+hypopnea index >= 10/hour
Groups:
- Total: Total of all reporting groups
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.9) | 58.3 (12.0) | 58.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 72 | 73 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 22 | 41
  White | 59 | 56 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 78 | 156
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — measure weight and height compute as kg divided by height squared
  kg/m^2 | 34.9 (6.0) | 34.2 (5.8) | 34.6 (5.9)
apnea+hypopnea index [Mean (Standard Deviation); unit: number of apneas and hypopneas /hour] — AHI from Home sleep apnea test
  number of apneas and hypopneas /hour | 31.0 (19.1) | 28.6 (18.2) | 29.8 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Positive Airway Pressure Adherence (Nightly Use of Treatment)
Description: average nightly hours of using positive airway pressure (including 0 for nights not used)
Time Frame: 6 weeks after starting treatment
Population: patients using cpap or apap at clinic visit
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Number analyzed (Participants) | 59 | 66
hours | 3.99 (2.3) | 4.45 (2.3)
Statistical Analysis 1: Comparison: PSG CPAP Titration Then CPAP Treatment vs Auto-Adjusting Positive Airway Pressure; Test type: Non-Inferiority or Equivalence — Non-inferiority margin -0.55 (mean hours of APAP arm no lower than 0.55 hours below CPAP arm); p = 0.27, t-test, 2 sided — level of significance <0.05, Power = 0.80; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-.35 to 1.26], Standard Error of Mean 0.40

2. Secondary Outcome: Change in Epworth Sleepiness Scale
Description: Epworth sleepiness scale (ESS) is measure of subjective sleepiness. Tendency to fall asleep in 8 situations. Total varies from zero to 24. A ESS of 10 or less is considered normal. The change in the ESS = post-treatment value - pre-treatment value. A decrease in the ESS (negative change) is consistent with less sleepiness.
Time Frame: 6 weeks after starting treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Number analyzed (Participants) | 59 | 66
units on a scale | -3.7 (4.8) | -4.1 (4.7)
Statistical Analysis 1: Comparison: PSG CPAP Titration Then CPAP Treatment vs Auto-Adjusting Positive Airway Pressure; Patients using PAP (average of >=1/2 hour per night) at 6 weeks clinic visit; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.3 to 2.1]

3. Secondary Outcome: Change in Functional Outcomes of Sleep Questionnaire
Description: The functional outcomes of sleep questionnaire (FOSQ) is a standard quality of life measure used to assess improvement in quality of life after treatment for sleep disorders. The total FOSQ score was analyzed. The range if 5 to 20. A higher score is a better quality of life. This analysis compares the change after treatment (post treatment FOSQ - pretreatment FOSQ). A positive difference indicates an improve in the quality of life.
Time Frame: 6 weeks at clinic
Population: Using PAP 1/2 hour or more nightly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Number analyzed (Participants) | 59 | 66
units on a scale | 2.2 (3.7) | 2.6 (3.5)
Statistical Analysis 1: Comparison: PSG CPAP Titration Then CPAP Treatment vs Auto-Adjusting Positive Airway Pressure; Patients using PAP (average >=1/2 hour per nightly use) at 6 weeks clinic visit; Test type: Superiority or Other; p = 0.33, t-test, 2 sided — < 0.05 criteria for statistical significance; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-0.73 to 2.1], Standard Error of Mean 0.71

4. Secondary Outcome: Residual Apnea-hypopnea Index
Description: The PAP device estimate of residual apnea-hypopnea index (AHI, number of apneas and hypopneas per hour of patient use) an estimate of effectiveness of treatment. An AHI < 10 is considered adequate treatment and <5/hour ideal treatment.
Time Frame: over first 6 weeks of treatment
Population: participants using PAP at clinic visit (>= 1/2 hour of nightly use)
Measure: Mean (Standard Deviation); unit: events (apneas+hypopneas)/hour
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Number analyzed (Participants) | 59 | 66
events (apneas+hypopneas)/hour | 4.9 (4.9) | 5.5 (4.7)
Statistical Analysis 1: Comparison: PSG CPAP Titration Then CPAP Treatment vs Auto-Adjusting Positive Airway Pressure; Patients using PAP (average >= 1/2 hour of nightly use) at 6 weeks clinic visit; Test type: Superiority or Other; p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-1.12 to 2.29]

5. Secondary Outcome: Treatment Pressure (Level of CPAP or 90th Percentile APAP)
Description: The level of CPAP used for treatment versus the 90th percentile pressure used during APAP. The 90th percentile pressure is the value that is used if one converts a patient from APAP to CPAP.
Time Frame: 6 weeks clinic
Population: participants using PAP at the 6 weeks clinic visit
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Number analyzed (Participants) | 59 | 66
cm H2O | 11.7 (2.5) | 10.8 (3.1)
Statistical Analysis 1: Comparison: PSG CPAP Titration Then CPAP Treatment vs Auto-Adjusting Positive Airway Pressure; participants using PAP (average >=1/2 hour of use) at 6 weeks clinic visit; Test type: Superiority or Other; p = 0.07, t-test, 2 sided — P < 0.05 considered statistically significant; Mean Difference (Final Values) = - 0.92, 95% CI 2-sided [-1.92 to 0.09], Standard Error of Mean 0.51

ADVERSE EVENTS:
Time Frame: Study duration
Arm/Group | PSG CPAP Titration Then CPAP Treatment | Auto-Adjusting Positive Airway Pressure
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 19/78 | 12/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSG CPAP Titration Then CPAP Treatment (N=78) | Auto-Adjusting Positive Airway Pressure (N=78)
PAP treatment intolerance (General disorders) | 19 (19) | 12 (12) — unable to use PAP

LIMITATIONS AND CAVEATS:
Carefully selected group with male predominance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No